CLINICAL TRIAL: NCT03642873
Title: A Study Designed to Examine the Potential for a Drug-drug Interaction Between Guaifenesin and Hydrocodone Bitartrate in Normal Healthy Volunteers
Brief Title: Study to Evaluate Drug-drug Interactions of Guaifenesin and Hydrocodone Bitartrate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 2006-HYDRO-04
Record Dates: First submitted 2018-08-20; First posted 2018-08-22 (Actual); Results first posted 2019-06-20 (Actual); Last update posted 2019-06-20 (Actual); Status verified 2019-03

CONDITIONS: Healthy Subjects
MeSH Terms: interventions — Guaifenesin; Hydrocodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Guaifenesin (Humibid®) single extended release 1200 mg tablet administered with 240 mL of room temperature water under fasted conditions.
  Interventions: Drug: Humibid®
- Treatment B (Experimental): Hydrocodone Bitartrate of 10 mg in 3 oral doses of a single 3.33 mg tablet in three intervals administered with 240 mL of room temperature water in the fasted state.
  Interventions: Drug: Hydrocodone Bitartrate
- Treatment C (Experimental): Hydrocodone Bitartrate 10 mg in 3 oral doses of a single 3.33 mg tablet in three intervals and guaifenesin (Humibid®) 1200 mg ER administered with 240 mL of room temperature water in the fasted state.
  Interventions: Drug: Humibid® and Hydrocodone Bitartrate tablet

INTERVENTIONS:
Drug: Humibid® — Humibid® 1200 mg (single extended release) tablet
  Other Names: Guaifenesin
  Arms: Treatment A
Drug: Hydrocodone Bitartrate — Hydrocodone Bitartrate (3.33 mg q4h X 3)
  Arms: Treatment B
Drug: Humibid® and Hydrocodone Bitartrate tablet — Humibid® 1200 mg (single extended release) tablet and Hydrocodone bitartrate (3.33 mg q4h X 3)
  Arms: Treatment C

SUMMARY:
Determine and compare the plasma concentrations and safety and tolerability of Guaifenesin and hydrocodone bitartrate when they are administered alone or in combination to normal healthy male and/or female subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and/or females between the ages of 19 and 55 years, inclusive.
2. Females of childbearing potential were using one of the following acceptable birth control methods:

   * Intrauterine device (IUD) in place for at least 3 months prior to study;
   * Barrier method (condom or diaphragm) with spermicide for at least 14 days prior to screening through 30 days beyond study completion;
   * Stable hormonal contraceptive for at least 3 months prior to study through 30 days beyond completion of study;

   Abstinence was not an acceptable form of contraception.

   Females of non-childbearing potential were surgically sterile (bilateral tubal ligation with surgery at least 6 months prior to study, hysterectomy, or bilateral oophorectomy at least 3 months prior to study) or postmenopausal <2 years. An FSH >40 mIU/mL was obtained and in the record.
3. Good general health was determined by medical history, physical examination, electrocardiogram (ECG), and clinical laboratory measures.
4. Within 15% of Ideal Body Weight as defined by the 1983 Metropolitan Life chart.
5. Non-tobacco users, who had not used nicotine or nicotine-containing products for at least 1 year.
6. Able to read, understand, and sign the informed consent after the nature of the study had been explained.
7. Negative finding on tests for Hepatitis B and C antigen as well as HIV and pregnancy test (if female).
8. Negative urine screen for drugs of abuse and alcohol at screening and the first check in.
9. Non-alcohol or drug abuser - for alcohol, defined as history of less then 4 drinks daily.

Exclusion Criteria:

1. Clinically significant abnormalities detected by medical history, physical, ECG, or clinical laboratory findings (as determined by the Principal Investigator). Any disease or condition which impacted absorption, distribution, metabolism, or elimination of the study drugs.
2. Females who were pregnant or nursing.
3. History of hypersensitivity reaction to the study drugs or related compounds, such as other opioids.
4. Receipt of an investigational drug within 1 month prior to study enrollment.
5. Donation of blood or significant loss of blood within 56 days or plasma within 14 days prior study enrollment.
6. Known or suspected use of illicit drugs (including codeine or hydrocodone, etc.).
7. The use of any medication on a chronic basis with the exception of oral contraceptives for women of childbearing potential. An appropriate drug-free period for prescription or over-the-counter (OTC) drugs provided to washout any especially long half-life drugs.
8. Consumption of alcohol within 48 hours prior to each dosing period.
9. Consumption of grapefruit 14 days prior to dosing and throughout the study.
10. Hemoglobin value < 12 g/dL. If a subject's hemoglobin dropped below 11.0 g/dL the subject was dropped from the study at the Principal Investigator's discretion.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-05-05 (Actual); Primary Completion 2007-05-21 (Actual); Study Completion 2007-05-21 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single-centre study.
Pre-assignment Details: A total of 24 subjects entered the study, among them 23 subjects completed the study.
Groups:
- Sequence ABC: First Intervention Treatment A: Single Humibid® 1200 mg guaifenesin Extended Release (ER) bi-layer tablet by mouth under fasted state
  Second Intervention Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Third Intervention Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
- Sequence ACB: First Intervention Treatment A: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
  Second Intervention Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Third Intervention Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
- Sequence BAC: First Intervention Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Second Intervention Treatment A: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
  Third Intervention Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
- Sequence BCA: First Intervention Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Second Intervention Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Third Intervention Treatment A: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
- Sequence CAB: First Intervention Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Second Intervention Treatment A: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
  Third Intervention Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
- Sequence CBA: First Intervention Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Second Intervention Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Third Intervention Treatment A: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
Period: First Intervention (1 Day)
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Intervention (1 Day)
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Washout (7 Days)
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 4 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Third Intervention (1 Day)
Arm/Group | Sequence ABC | Sequence ACB | Sequence BAC | Sequence BCA | Sequence CAB | Sequence CBA
Started | 4 | 4 | 4 | 4 | 4 | 4
Completed | 4 | 4 | 4 | 4 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Screen failure | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants were randomized at each visit to receive either
  Treatment A (Reference): Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
  Treatment B (Reference): Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Treatment C (Test): Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
  Scheduled Washout of 7 days between each doses.
  All study participants received all three treatments
Arm/Group | All Study Participants
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 29.6 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian | 1
  Asian | 1
  Black | 2
  Caucasian | 17
  Hispanic | 3
Weight [Mean (Standard Deviation); unit: lb] | 148.3 (18.8)
Height [Mean (Standard Deviation); unit: Inches] | 67.5 (3.3)
Elbow Breadth [Mean (Standard Deviation); unit: Inches] | 2.6 (0.2)
Frame Size [Number; unit: participants]
  Small | 7
  Medium | 15
  Large | 2

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Guaifenesin
Description: Pharmacokinetic Parameter Cmax (Maximum measured plasma concentration)
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 11, 13, 16, 20, 24, and 26 hours Post dose
Population: Pharmacokinetic (PK) Data Sets included all the 24 subjects for analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Treatment A (Reference) - Plasma Guaifenesin: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state.
- Treatment C (Test) - Plasma Guaifenesin; Treatment C (Test) - Plasma Hydrocodone Bitartrate: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state.
- Treatments B (Reference) - Plasma Hydrocodone Bitartrate: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state.
Arm/Group | Treatment A (Reference) - Plasma Guaifenesin | Treatment C (Test) - Plasma Guaifenesin | Treatments B (Reference) - Plasma Hydrocodone Bitartrate | Treatment C (Test) - Plasma Hydrocodone Bitartrate
Number analyzed (Participants) | 24 | 24 | 23 | 24
ng/mL | 1770 (628) | 1810 (784) | 11.3 (2.14) | 11.3 (1.78)

2. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to the Last Measurable Concentration (AUC(0-t)) of Guaifenesin
Description: Pharmacokinetic Parameter AUC(0-t) The area under the plasma concentration versus time curve from time 0 to time of the last measurable concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 11, 13, 16, 20, 24, and 26 hours Post dose
Population: Pharmacokinetic (PK) Data Sets
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A (Reference) - Plasma Guaifenesin | Treatment C (Test) - Plasma Guaifenesin | Treatments B (Reference) - Plasma Hydrocodone Bitartrate | Treatment C (Test) - Plasma Hydrocodone Bitartrate
Number analyzed (Participants) | 24 | 24 | 23 | 24
ng*hr/mL | 8286.2 (2440.0) | 8186.7 (2801.0) | 133.36 (29.407) | 132.99 (23.053)

3. Primary Outcome: Area Under Plasma Concentration-time Curve From Time 0 to Infinity (AUC(0-inf)) of Guaifenesin
Description: The area under the plasma concentration versus time curve from time 0 to infinity, calculated as AUC(0-t) + Ct/ Kel, where Ct is the last measurable concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 11, 13, 16, 20, 24, and 26 hours Post dose
Population: Pharmacokinetic (PK) Data Sets
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Treatment A (Reference) - Plasma Guaifenesin | Treatment C (Test) - Plasma Guaifenesin | Treatments B (Reference) - Plasma Hydrocodone Bitartrate | Treatment C (Test) - Plasma Hydrocodone Bitartrate
Number analyzed (Participants) | 20 | 21 | 23 | 24
ng*hr/mL | 8501.5 (2784.5) | 8347.8 (2762.4) | 140.44 (32.792) | 139.70 (26.044)

4. Primary Outcome: Apparent Terminal Elimination Rate Constant (Kel) of Guaifenesin
Description: Apparent first-order terminal elimination rate constant calculated from a semi-log plot of the plasma concentration versus time curve. The parameter was calculated by linear least-squares regression analysis using the maximum number of points in the terminal log-linear phase.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 11, 13, 16, 20, 24, and 26 hours Post dose
Population: Pharmacokinetic (PK) Data Sets
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | Treatment A (Reference) - Plasma Guaifenesin | Treatment C (Test) - Plasma Guaifenesin | Treatments B (Reference) - Plasma Hydrocodone Bitartrate | Treatment C (Test) - Plasma Hydrocodone Bitartrate
Number analyzed (Participants) | 20 | 21 | 23 | 24
1/hr | 0.205 (0.104) | 0.207 (0.199) | 0.151 (0.0251) | 0.155 (0.0233)

5. Primary Outcome: Time to Maximum Observed Concentration (Tmax) of Guaifenesin
Description: Pharmacokinetic Parameter (Tmax) Time of the maximum measured plasma concentration.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 11, 13, 16, 20, 24, and 26 hours Post dose
Population: Pharmacokinetic (PK) Data Sets
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A (Reference) - Plasma Guaifenesin | Treatment C (Test) - Plasma Guaifenesin | Treatments B (Reference) - Plasma Hydrocodone Bitartrate | Treatment C (Test) - Plasma Hydrocodone Bitartrate
Number analyzed (Participants) | 24 | 24 | 23 | 24
hr | 1.08 (0.551) | 1.04 (0.415) | 9.59 (2.16) | 9.33 (2.09)

6. Primary Outcome: Apparent Terminal Elimination Half-life (T1/2) of Guaifenesin
Description: Apparent first-order terminal elimination half-life was calculated as 0.693/Kel.
Time Frame: 0 (pre-dose), 0.5, 1, 1.5, 2, 3, 4, 4.5, 5, 5.5, 6, 7, 8, 8.5, 9, 9.5, 10, 11, 13, 16, 20, 24, and 26 hours Post dose
Population: Pharmacokinetic (PK) Data Sets
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Treatment A (Reference) - Plasma Guaifenesin | Treatment C (Test) - Plasma Guaifenesin | Treatments B (Reference) - Plasma Hydrocodone Bitartrate | Treatment C (Test) - Plasma Hydrocodone Bitartrate
Number analyzed (Participants) | 20 | 21 | 23 | 24
hr | 4.82 (3.30) | 5.34 (3.13) | 4.71 (0.833) | 4.60 (0.831)

7. Secondary Outcome: Number of Adverse Events(AEs) Experienced by Participants
Description: Intensity was determined by the Investigator. For symptomatic AEs the following definitions were applied.
  Mild = AE did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/ pain.
  Relationship to Investigational Medicinal Products (IMP) Unlikely = Slight, but remote, chance that AE was caused by IMP. Possible = Reasonable suspicion that the AE was caused by IMP. Probable = Most likely that AE was caused by IMP.
Time Frame: Upto Day 17
Population: Pharmacokinetic (PK) Data Sets
Measure: Number; unit: Events
Groups:
- Treatment A: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet by mouth under fasted state
- Treatment B: Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
- Treatment C: Single Humibid® 1200 mg guaifenesin Extended-Release (ER) bi-layer tablet and Hydrocodone Bitartrate 10 mg (3.33 mg q4h X 3) tablet by mouth under fasted state
Arm/Group | Treatment A | Treatment B | Treatment C
Number analyzed (Participants) | 24 | 23 | 24
Events
  TEAE by severity: Mild | 7 | 12 | 25
  TEAE by severity: Moderate | 0 | 1 | 0
  TEAE by severity: Severe | 0 | 0 | 0
  Relationship to IMP - Unlikely | 4 | 0 | 1
  Relationship to IMP - Possible | 3 | 8 | 8
  Relationship to IMP - Probable | 0 | 5 | 16

ADVERSE EVENTS:
Time Frame: Up to Day 17
Arm/Group | Treatment A | Treatment B | Treatment C
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/23 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 5/24 | 10/23 | 10/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment A (N=24) | Treatment B (N=23) | Treatment C (N=24)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Lacrimation increased (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 4 (4) | 2 (2)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Clumsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 6 (8)
Head discomfort (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 5 (5) | 5 (6)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No